CLINICAL TRIAL: NCT06313060
Title: Efficacy of Carbonated Beverages in the Resolution of Alimentary Esophageal Impaction: a Multicenter Randomized Clinical Trial
Brief Title: Efficacy of Carbonated Beverages in the Resolution of Alimentary Esophageal Impaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, Marina de Benito Sanz, Principal investigator, Hospital del Rio Hortega
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 010
Record Dates: First submitted 2024-03-02; First posted 2024-03-15 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Esophagus Disorder
MeSH Terms: conditions — Esophageal Diseases

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 200 ml of Coca-Cola will be administered and must be ingested within a maximum of 10 minutes
  Interventions: Dietary Supplement: Coca-cola
- Control group (No Intervention): will not receive any type of medication or drink

INTERVENTIONS:
Dietary Supplement: Coca-cola — 200 ml of Coca-Cola will be administered and must be ingested within a maximum of 10 minutes
  Arms: Intervention group

SUMMARY:
Objectives: To evaluate the efficacy of the administration of carbonated beverages in the resolution of dietary esophageal impaction, and to identify subgroups in which their effectiveness may be different: patients with/without esophageal diseases, with/without a history of impaction.

Methods: A clinical trial was conducted randomizing consecutive patients with a clinical diagnosis of dietary esophageal impaction to receive 200cc of carbonated drink or not at all, excluding patients with a previous diagnosis of non-esophageal stenosis that could not be overcome with a gastroscope and suspected impaction by non-alimentary foreign bodies, spines or bones. Subsequently, an endoscopic evaluation will be carried out in all cases, checking the presence or absence of a foreign body and removing it if necessary, as well as assessing and recording the possible underlying esophageal pathology.

A telephone follow-up will be carried out after 7 days, recording possible adverse events.

DETAILED DESCRIPTION:
METHODOLOGY

1. Design: Randomized multicenter clinical trial.
2. Period: patients treated in the Emergency Department with a clinical diagnosis of esophageal foreign body impaction (cervical or retrosternal foreign body sensation, hypersalivation, inability to swallow) will be collected with indication by clinical practice by the emergency physician who evaluates them for upper gastrointestinal endoscopy.
3. Population selection:

   * Scope: patients treated in the Emergency Department of the participating hospitals.
   * Inclusion and exclusion criteria:

     * The inclusion criteria are:
     * Patients who come to the Emergency Department with a clinical diagnosis of esophageal impaction due to food bolus (determined by at least one of the following symptoms: sialorrhea, inability to swallow or cervical or retrosternal foreign body sensation) that requires endoscopic extraction.
     * Age greater than or equal to 18 years of age. The inclusion criterion related to age refers to the age at the date of signing the informed consent form.
     * The exclusion criteria are:
     * Pregnancy.
     * Benign or malignant esophageal stricture that cannot be overcome with a conventional gastroscope.
     * Patients with intraesophageal prostheses
     * Non-food foreign body (includes fish bones or bones)
     * Ingestion of some type of carbonated beverage after impaction.
     * Contraindication for the administration of carbonated drink (Cola-Cola) due to allergy or intolerance to any of its components.

   3.3. Recruitment procedure: all patients treated in the Emergency Department of the aforementioned hospitals with a clinical diagnosis of esophageal food impaction who meet the inclusion criteria and do not meet the exclusion criteria will be invited by the Emergency Department to participate in the study.

   3.4. Sample size Most of the studies on carbonated beverages date from the 1980s and 1990s, are very short series, and in some of them they are combined with the administration of glucagon. In all of them, the success rate is 100%.

   In the largest and most recent series of the studies reviewed, the effectiveness rate of the carbonated drink is 59%, which in the light of clinical experience may be exaggerated (possible bias in the selection of the most favorable patients). If no treatment is performed, the foreign body can be found in 80-90% of cases. Thus, considering a difference of 20% relevant, assuming a success rate in the intervention group of 35%, with a risk α=5% and a power of 80%, a total of 84 patients per group would be needed. Since the study has no follow-up, we consider it unlikely that there will be any losses.

   In light of the results of our placebo-controlled clinical trial on the efficacy of glucagon, in which the only difference detected was a decrease in the complexity of endoscopy in the intervention group in patients with no personal history of impaction, it would be interesting to have a number of such patients in order to be able to detect differences with adequate power. According to our study, 47% of patients (66/140) have no history of impaction that required medical assistance. Thus, if we consider the n properly calculated as patients with no history, we need a total of 177 patients per group.
4. Intervention 4.1. Randomization It will be carried out once the patient agrees to participate in the work and the absence of exclusion criteria is verified. A stratified randomization will be carried out by center, so that each participating center will have its sealed randomization sequence. Within each stratum, pure randomization will be performed using a computer-generated sequence where the probability of belonging to each group will be 0.5. A total of 100 numbered opaque sealed envelopes will be available for each centre and will be stored in the emergency department and opened consecutively as patients are included.

   4.2. Intervention The study will be completed after the formalization of the informed consent in accordance with Law 41/2002 on patient autonomy. Participation in the study will not alter your relationship with your doctor.

   4.2.1 Pre-endoscopic evaluation

   Patients will be identified in the emergency department. Those who meet the inclusion criteria and do not present any exclusion criteria will be invited to participate in the study. Once they consent to their participation, the endoscopist on duty will be contacted to plan the examination, which should be carried out in 30-120 minutes after the call in both groups. Once the endoscopic examination has been scheduled, the patient will be randomized. Based on this, 2 groups are established:
   * Intervention group: 200 ml of Coca-Cola will be administered and must be ingested within a maximum of 10 minutes.
   * Control group: You will not receive any type of medication or drink. 4.2.3 Endoscopic evaluation The endoscopic examination should be performed at least 30 minutes after the administration of the drink and within 2 hours of the call. In the control group, endoscopy will be performed between 30 and 120 minutes after the call. It will be carried out according to the usual protocols in each center. The presence or absence of foreign bodies, the maneuvers for their extraction, and the underlying esophageal findings will be collected in the endoscopic report in a systematic manner. The decision about which interventions to perform if the presence of the foreign body is documented is in the hands of the endoscopist who performs the examination.
5. Data collection 5.1 Description of variables

   * Effect: Patients in whom the endoscopic examination does not show an image of an impacted foreign body in the esophagus will be considered a success. Patients in whom an impacted foreign body is endoscopically documented will be considered a therapeutic failure.
   * Impacted foreign body: It is defined as any mass, regardless of its origin, that is fixed, without the ability to mobilize spontaneously, at some point in the esophagus. It is opposed to the non-impacted foreign body, the one that is in the esophagus but mobilizes spontaneously, without requiring any type of endoscopic maneuver.
   * The difficulty of the examination will be measured indirectly with the following variables:
   * Duration of the scan: Time interval (in minutes) from the time the endoscope is inserted to the time it is removed.
   * Duration of extraction: In patients in whom a foreign body is identified, the time interval (in minutes) from the time the first tool is inserted to attempt extraction (or, if the attempt is made to advance to the gastric chamber using the endoscope from the first attempt to mobilize the foreign body) until the foreign body is removed from its position.

   5.2. Data sources Variable variables related to the patient's personal history will be collected in the form of an interview with the patient by the emergency physician, focusing on the presence of esophageal pathology, medications that affect esophageal motility and history of impactions, time of impaction and water intake after obstruction.

   After performing the endoscopy, the physician who performs it will collect technical details such as the endoscopy time, the tools used for deimpaction, the type and location of the foreign body and the underlying esophageal pathology 5.3. Existence of a blind person It is not possible to conduct a double-blind study as the intervention (administration of carbonated beverage) cannot be compared with placebo. Patients in the Emergency Department will be instructed not to disclose to the endoscopist to which branch of the study they have been assigned.

   Although the final report to be delivered to the patient at hospital discharge will include the treatment administered, since it is generated and delivered to the patient after the procedure has been performed. The evaluation of the efficacy of the treatment will be performed by the endoscopist during the endoscopic examination. Since the endoscopy unit does not have access to the software or treatment sheets of the emergency department, the endoscopists in charge of evaluating the outcome of the treatment will not be able to know the assigned group.
6. Follow-up 7-10 days after the endoscopic examination, a standardized telephone interview will be conducted to assess the possible presence of adverse effects. In case of the presence of symptoms, the causal relationship with the procedure will be evaluated by a group of 3 study investigators. The severity of the events will be assessed according to the usual classifications (CTCAE v.4) and according to the definitions of Royal Decree 1090/2015.
7. Analysis The statistical analysis of these will be carried out using the STATA program (StataCorp. Version 16. Stata Statistical Software. College Station, TX).

   To verify that there are no imbalances between the experimental group and the control, means are compared with quantitative variables, assessing the magnitude of the association with Pearson's correlation coefficient (r). For binary categorical variables, proportions are compared, assessing the association with the OR obtained by logistic regression. For ordinal categoricals, the ROs are calculated with respect to the category determined as a reference.

   For the descriptive variables, the arithmetic mean and the standard deviation will be calculated for the quantitative variables (variables that do not follow a normal distribution according to the Kolmogorov-Smirnov test will be described with median, minimum, maximum and interquartile range), and the qualitative variables will be expressed as percentages and their 95% confidence intervals.

   The analysis of the primary endpoint, the proportion of patients without the presence of an impacted foreign body in both groups, will be compared using the homogeneity z-test without using the Yates correction. The confidence interval of the difference between the two groups will also be estimated. The analysis will be performed on an intention-to-treat basis and on a per-protocol basis (including only subjects who receive treatment within and perform the examination within the predetermined time frames).

   Within the secondary endpoints, the proportion of complications in both groups will be checked by the χ2 test. The duration of the procedures will be compared using the Student's t-test. Multivariate logistic regression techniques will be used to evaluate the factors associated with the effectiveness of the treatment.
8. Novelty, originality This study continues a line of research established at our center with a previous clinical trial on the efficacy of glucagon with a sample size and a novel design, which provides data not demonstrated in randomized trials.

The efficacy of carbonated beverages for this indication has also not been proven with a study of the characteristics of the one we propose. Our findings would avoid unnecessary endoscopies, if the efficacy of these beverages is demonstrated, including them in the protocol of action in food esophageal impaction. Or, if, on the contrary, it were to prove ineffective, unnecessary waiting for endoscopy and inconvenience to the patient when attempting these futile measures would be avoided.

ELIGIBILITY:
Inclusion Criteria:

* -Patients who come to the Emergency Department with a clinical diagnosis of esophageal impaction due to food bolus (determined by at least one of the following symptoms: sialorrhea, inability to swallow or cervical or retrosternal foreign body sensation) that requires endoscopic extraction.
* Age greater than or equal to 18 years of age. The inclusion criterion related to age refers to the age at the date of signing the informed consent form.

Exclusion Criteria:

* -Pregnancy.
* Benign or malignant esophageal stricture that cannot be overcome with a conventional gastroscope.
* Patients with intraesophageal prostheses
* Non-food foreign body (includes fish bones or bones)
* Ingestion of some type of carbonated beverage after impaction.
* Contraindication for the administration of carbonated drink (Cola-Cola) due to allergy or intolerance to any of its components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of carbonated beverage for disimpaction | 3 years
  Number of patients with esophageal impaction resolved with the carbonated beverage

CONTACTS AND LOCATIONS:
Locations (1):
- Manuel Perez-Miranda, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No